CLINICAL TRIAL: NCT00875017
Title: An Open-label, Phase I, One-dose, One-meal, Balance Study Comparing the Absorption of Dietary Phosphorus When Administering FOSRENOL® (Lanthanum Carbonate) or RENVELA® (Sevelamer Carbonate) in Healthy Adult Volunteers
Brief Title: Comparing Absorption of Dietary Phosphorus When Administering FOSRENOL® or RENVELA® in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SPD405-128
Record Dates: First submitted 2009-01-22; First posted 2009-04-03 (Estimated); Results first posted 2010-07-02 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Meal + Lanthanum (Experimental)
  Interventions: Drug: Lanthanum Carbonate
- Meal + Sevelamer (Active Comparator)
  Interventions: Drug: Sevelamer
- Meal Only (No Intervention)
- Fasting (No Intervention)

INTERVENTIONS:
Drug: Lanthanum Carbonate — 1 x 1000mg tablet
  Other Names: Fosrenol
  Arms: Meal + Lanthanum
Drug: Sevelamer — 3 x 800mg tablets
  Other Names: Renvela
  Arms: Meal + Sevelamer

SUMMARY:
The purpose of this study is to compare the absorption of dietary phosphorus following a single dose with lanthanum carbonate (1000mg) and a single dose of sevelamer carbonate (2400mg).

ELIGIBILITY:
Inclusion Criteria

* Ability to provide informed consent to participate in the study.
* Healthy volunteers, age 19-45 inclusive.
* Subject must be willing to comply with applicable contraceptive requirements of the protocol
* Female subjects must have a negative pregnancy test
* Satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination, vital signs, ECG and laboratory evaluation.
* Body Mass Index (BMI) between 20.0 and 29.9kg/m² inclusive.
* Serum 1.25 dihydroxy vitamin D3 >30pg/mL.
* Ability to chew or swallow a dose of the investigational products and mannitol solution as prescribed in the protocol.
* Ability and willingness to fast for up to 24 hours.

Exclusion Criteria

* Current or recurrent disease that could affect the action, absorption or disposition of the investigational products utilized in this study, or could affect clinical or laboratory assessments.
* Current or relevant previous history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or study procedures.
* Significant illness within 2 weeks of the first dose of investigational product.
* Current use of any medication with the exception of hormonal replacement therapy or hormonal contraceptives within 14 days of first dose of investigational product.
* Known or suspected intolerance or hypersensitivity to the investigational product(s) or mannitol solution, closely related compounds or any of the stated ingredients.
* History of alcohol or other substance abuse within the last year.
* A positive screen for alcohol or drugs of abuse.
* Male subjects who consume more than 21 units of alcohol per week or three units per day. Female subjects who consume more than 14 units of alcohol per week or two units per day.
* A positive human immunodeficiency virus (HIV) antibody screen, Hepatitis B surface antigen (HBsAg) or Hepatitis C virus (HCV) antibody screen.
* Use of tobacco in any form or other nicotine-containing products in any form. Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the first dose of investigational product.
* Routine consumption of more than two units of caffeine per day or subjects who experience caffeine withdrawal headaches.
* Donation of blood or blood products within 60 days prior to receiving the first dose of investigational product.
* Use of another investigational product within 30 days prior to receiving the first dose of investigational product or active enrolment in another drug or vaccine clinical study.
* An inability to follow a standardized diet and/or meal schedule, as required during the study.
* Substantial changes in eating habits within 30 days prior to receiving the first dose of investigational product, as assessed by the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04-20 (Actual); Primary Completion 2009-06-16 (Actual); Study Completion 2009-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States

REFERENCES:
- [Result] Martin P, Wang P, Robinson A, Poole L, Dragone J, Smyth M, Pratt R. Comparison of dietary phosphate absorption after single doses of lanthanum carbonate and sevelamer carbonate in healthy volunteers: a balance study. Am J Kidney Dis. 2011 May;57(5):700-6. doi: 10.1053/j.ajkd.2010.11.028. Epub 2011 Feb 26. PMID 21354682
- [Result] Behets GJ, Dams G, Damment SJ, Martin P, De Broe ME, D'Haese PC. Differences in gastrointestinal calcium absorption after the ingestion of calcium-free phosphate binders. Am J Physiol Renal Physiol. 2014 Jan 1;306(1):F61-7. doi: 10.1152/ajprenal.00219.2013. Epub 2013 Nov 6. PMID 24197066
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized to one of 6 treatment sequences each of which consisted of four treatment periods separated by a 7-14 day washout period. In each of the first three treatment periods subjects received lanthanum carbonate 100mg +meal, sevelamer carbonate 2400mg+meal or meal. Subjects fasted in the fourth treatment period.
Groups:
- Sequence 1: Lanthanum carbonate (1000 mg) + meal in first intervention period, washout, Sevelamer carbonate (2400 mg) + meal in second intervention period, washout, Meal only in third intervention period, washout, Fasting in fourth intervention period
- Sequence 2: Sevelamer carbonate (2400 mg) + meal in first intervention period, washout, Meal only in second intervention period, washout, Lanthanum carbonate (1000 mg) + meal in third intervention period, washout, Fasting in fourth intervention period
- Sequence 3: Meal only in first intervention period, washout, Lanthanum carbonate (1000 mg) + meal in second intervention period, washout, Sevelamer carbonate (2400 mg) + meal in third intervention period, washout, Fasting in fourth intervention period
- Sequence 4: Lanthanum carbonate (1000 mg) + meal in first intervention period, washout, Meal only in second intervention period, washout, Sevelamer carbonate (2400 mg) + meal in third intervention period, washout, Fasting in fourth intervention period
- Sequence 5: Sevelamer carbonate (2400 mg) + meal in first intervention period, washout, Lanthanum carbonate (1000 mg) + meal in second intervention period, washout, Meal only in third intervention period, washout, Fasting in fourth intervention period
- Sequence 6: Meal only in first intervention period, washout, Sevelamer carbonate (2400 mg) + meal in second intervention period, washout, Lanthanum carbonate (1000 mg) + meal in third intervention period, washout, Fasting in fourth intervention period
Period: First Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 5 | 5 | 5 | 6 | 5 | 5
Completed | 3 | 5 | 4 | 5 | 4 | 5
Not Completed | 2 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Problems collecting rectal effluent | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Intolerance to nasogastric tube | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 5 | 4 | 5 | 4 | 5
Completed | 3 | 5 | 3 | 5 | 4 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Problem collecting rectal effluent | 0 | 0 | 1 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 5 | 3 | 5 | 4 | 5
Completed | 3 | 5 | 3 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 5 | 3 | 4 | 4 | 5
Completed | 3 | 4 | 3 | 4 | 4 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Problems collecting rectal effluent | 0 | 1 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 4 | 3 | 4 | 4 | 5
Completed | 3 | 3 | 2 | 4 | 4 | 5
Not Completed | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 2 | 4 | 4 | 5
Completed | 3 | 3 | 2 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Fourth Intervention
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 3 | 3 | 2 | 4 | 3 | 5
Completed | 3 | 3 | 2 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Inability to comply with fasting | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 5 | 5 | 28
Age, Categorical [Count of Participants; unit: Participants] — Although 31 subjects were randomized in the study, the demographics are presented from the Safety Set (n = 28). Safety Set consisted of subjects who had at least one dose of investigational medicinal product and had at least one post-dose safety assessment.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 5 | 5 | 5 | 5 | 5 | 28
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Although 31 subjects were randomized in the study, the demographics are presented from the Safety Set (n = 28). Safety Set consisted of subjects who had at least one dose of investigational medicinal product and had at least one post-dose safety assessment.
  years | 26.0 (9.54) | 23.6 (2.07) | 24.4 (3.85) | 27.4 (9.71) | 25.8 (5.45) | 28.2 (6.38) | 25.9 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Although 31 subjects were randomized in the study, the demographics are presented from the Safety Set (n = 28). Safety Set consisted of subjects who had at least one dose of investigational medicinal product and had at least one post-dose safety assessment.
  Participants
    Female | 1 | 0 | 1 | 2 | 2 | 2 | 8
    Male | 2 | 5 | 4 | 3 | 3 | 3 | 20
Region of Enrollment [Count of Participants; unit: Participants] — Although 31 subjects were randomized in the study, the demographics are presented from the Safety Set (n = 28). Safety Set consisted of subjects who had at least one dose of investigational medicinal product and had at least one post-dose safety assessment.
  Participants
    United States | 3 | 5 | 5 | 5 | 5 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Net Phosphorous Absorption
Description: Net phosphorous absorption (Lanthanum carbonate period) = phosphorous ingested in meal minus (Rectal effluent phosphorous after Lanthanum carbonate + meal minus Rectal effluent phosphorous after fasting). Net phosphorous absorption (Sevelamer Carbonate period) = Phosphorous ingested in meal minus (Rectal effluent phosphorous after Sevelamer carbonate + meal minus Rectal effluent phosphorous after fasting). Net phosphorous absorption (Meal only period) = Phosphorous ingested in meal minus (Rectal effluent phosphorous after meal only minus Rectal effluent phosphorous after fasting).
Time Frame: 10 hours post-dose
Population: Pharmacodynamic Set (PD) consists of subjects who provided all rectal effluent collections and completed all treatment periods. Subjects who vomited during any of the treatment periods were excluded from the PD set.
Measure: Least Squares Mean (Standard Error); unit: mg
Groups:
- Lanthanum Carbonate: A meal containing a known amount of phosphorous is ingested along with oral administration of the phosphorous binder, lanthanum carbonate. 10 hours post-dose, rectal effluent is collected and the amount of phosphorous is measured.
- Sevelamer Carbonate: A meal containing a known amount of phosphorous is ingested along wuith oral administration of the phosphorous binder, sevelamer carbonate. 10 hours post-dose, rectal effluent is collected and the amount of phosphorous is measured.
- Meal Only: A meal containing a known amount of phosphorous is ingested. No phosphorous binder is administered. 10 hours post-meal, rectal effluent is collected and the amount of phosphorous is measured.
Arm/Group | Lanthanum Carbonate | Sevelamer Carbonate | Meal Only
Number analyzed (Participants) | 18 | 18 | 18
mg | 156.03 (14.161) | 221.78 (14.112) | 281.68 (14.112)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Sevelamer Carbonate; Net phosphorus absorption was analysed using a mixed linear effect model with fixed effects for sequence group, period and treatment group. Subject within sequence effect was included as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least Squares (LS) Mean Difference = -65.75, 95% CI [-96.01 to -35.49]
Statistical Analysis 2: Comparison: Lanthanum Carbonate vs Meal Only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -125.65, 95% CI [-155.91 to -95.39]
Statistical Analysis 3: Comparison: Sevelamer Carbonate vs Meal Only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -59.90, 95% CI [-89.87 to -29.93]

2. Secondary Outcome: Net Phosphorous Binding
Description: Net Phosphorous Binding (Lanthanum carbonate period) = Rectal effluent phosphorous after Lanthanum carbonate + meal minus Rectal effluent phosphorous after meal only. Net Phosphorous Binding (Sevelamer carbonate period) = Rectal effluent phosphorous after Sevelamer carbonate + meal minus Rectal effluent phosphorous after meal only.
Time Frame: 10 hours post-dose
Population: PD set
Measure: Least Squares Mean (Standard Error); unit: mg
Groups:
- Sevelamer Carbonate: A meal containing a known amount of phosphorous is ingested along with oral administration of the phosphorous binder, sevelamer carbonate. 10 hours post-dose, rectal effluent is collected and the amount of phosphorous is measured.
Arm/Group | Lanthanum Carbonate | Sevelamer Carbonate
Number analyzed (Participants) | 18 | 18
mg | 135.05 (12.348) | 63.15 (12.348)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Sevelamer Carbonate; Phosphorus binding was analysed using a mixed linear effect model with fixed effects for sequence group, period and treatment group. Subject within sequence effect was included as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = 71.90, 95% CI [40.03 to 103.77]

3. Secondary Outcome: Net Calcium Absorption
Description: Net Calcium Absorption (Lanthanum carbonate period) = Calcium ingested in meal minus (Rectal effluent calcium after Lanthanum carbonate + meal minus Rectal effluent calcium after fasting). Net Calcium Absorption (Sevelamer Carbonate period) = Calcium ingested in meal minus (Rectal effluent calcium after Sevelamer carbonate + meal minus Rectal effluent calcium after fasting). Net Calcium Absorption (Meal only period) = Calcium ingested in meal minus (Rectal effluent calcium after meal only minus Rectal effluent calcium after fasting).
Time Frame: 10 hours post-dose
Population: PD set
Measure: Least Squares Mean (Standard Error); unit: mg
Groups:
- Lanthanum Carbonate: A meal containing a known amount of calcium is ingested along with oral administration of the phosphorous binder, lanthanum carbonate. 10 hours post-dose, rectal effluent is collected and the amount of calcium is measured.
- Sevelamer Carbonate: A meal containing a known amount of calcium is ingested along with oral administration of the phosphorous binder, sevelamer carbonate. 10 hours post-dose, rectal effluent is collected and the amount of calcium is measured.
- Meal Only: A meal containing a known amount of calcium is ingested. No phosphorous binder is administered. 10 hours post-meal, rectal effluent is collected and the amount of calcium is measured.
Arm/Group | Lanthanum Carbonate | Sevelamer Carbonate | Meal Only
Number analyzed (Participants) | 18 | 18 | 18
mg | 49.46 (10.480) | 70.13 (10.450) | 65.02 (10.450)
Statistical Analysis 1: Comparison: Lanthanum Carbonate vs Sevelamer Carbonate; Net calcium absorption was analysed using a mixed linear effect model with fixed effects for sequence group, period and treatment group. Subject within sequence effect was included as a random effect; Test type: Superiority or Other; p = 0.049, Mixed Models Analysis; LS Mean Difference = -20.67, 95% CI [-41.22 to -0.13]
Statistical Analysis 2: Comparison: Lanthanum Carbonate vs Meal Only; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis; LS Mean Difference = -15.56, 95% CI [-36.11 to 4.99]
Statistical Analysis 3: Comparison: Sevelamer Carbonate vs Meal Only; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.612, Mixed Models Analysis; LS Mean Difference = 5.11, 95% CI [-15.24 to 25.47]

ADVERSE EVENTS:
Description: Due to the crossover design of the study, discontinuations during the course of the study will affect the number of subjects receiving each treatment. Therefore, the number of subjects for each treatment will be less than 28 (the total number of subjects in the Safety Set).
Arm/Group | Lanthanum Carbonate | Sevelamer Carbonate | Meal Only | Fasting
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/26 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 3/26 | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate (N=23) | Sevelamer Carbonate (N=24) | Meal Only (N=26) | Fasting (N=20)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.